CLINICAL TRIAL: NCT02629978
Title: Efficacy and Safety of Radiofrequency Ablation of Malignant Pulmonary Nodules
Brief Title: Radiofrequency Ablation of Malignant Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yueyong Xiao, Director of the Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-YY-006
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms; Carcinoma
Keywords: pulmonary; lung; cancer; carcinoma; nodule; malignant; radiofrequency ablation; RFA
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiofrequency ablation (Experimental): In this group, patients willingly receive CT-guided percutaneous radiofrequency ablation procedures are selected according to the inclusion criteria as follows. After a series of preoperative evaluation and preoperative preparation，the procedures will be performed under the CT guidance. CT/MRI scans will be ordered after 24-48 hours to see if there are complications (such as haemorrhage, pneumothorax and pleural effusion). Regularly follow-up will be carried out for several years after RFA to assess the effectiveness and safety of RFA integratedly.
  Interventions: Procedure: CT-guided percutaneous radiofrequency ablation

INTERVENTIONS:
Procedure: CT-guided percutaneous radiofrequency ablation — Percutaneous radiofrequency ablation (RFA) is a minimally invasive technique will be performed in patients with malignant pulmonary nodules in this group. RFA kills the tumors by causing coagulation necrosis via tissue heating. The electrode delivers thermal energy will be inserted into the target tissues under the CT guidance to ensure the area of ablation should cover the targets and the lung tissues 0.5-1.0 cm around the tumors. Post-operative scan and laboratory test will be conducted in time.
  Other Names: CT-guided percutaneous RFA

SUMMARY:
The objective of this study is to evaluate the outcomes of radiofrequency ablation in the treatment of patients with malignant pulmonary nodules（not exceed 3cm ）who are not suitable candidates for or refuse surgical resection.

DETAILED DESCRIPTION:
Percutaneous radiofrequency ablation (RFA) is a minimally invasive technique widely used to treat solid tumors. Patients with malignant pulmonary nodules will undergo a series of CT- guided percutaneous RFA procedures. During the procedures，percutaneous needles will be inserted into the target tissues under CT guidance，the needles deliver thermal energy and then destroy the tumors by causing coagulation necrosis via tissue heating. The purpose of this study is to assess the effectiveness and safety of RFA in pulmonary nodules （maximum tumor diameter ≦30 mm） was 10 mm apart from the big trachea, primary bronchi, esophagus, great vessels，heart and pleura. Preoperative and postoperative evaluations，including recent laboratory tests evaluated and imaging studies reviewed，will be performed both before and after the procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant pulmonary nodules.
2. Patients refuse or are not suitable for surgical resections.
3. 1-3 pulmonary nodules , with a maximum tumor diameter ≦30 mm.
4. Minimum distance of nodules are at least 10 mm apart from the surrounding tissues as big trachea, primary bronchi, esophagus, great vessels，heart and pleura.

Exclusion Criteria:

1. Patients who has uncorrectable coagulation disorders, severe heart or pulmonary failure, or uncontrolled infections.
2. With extensive extrapulmonary or intrapulmonary metastasis.
3. Have taken anticoagulant as aspirin in one week.
4. Target nodules nearby pleura or other important hilum and mediastinum structures.
5. With metal implants are adjacent to the target tissues which will be covered with ablation area.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
1- , 3- and 5-year survival rates | up to 5 years after the procedures
complication rate | During the procedure or up to 5 years after the procedures
  Including puncture-related complications such as pulmonary haemorrhage, hemothorax, pneumothorax, cardiac tamponade, and air embolism and ablation-related complications such as chest pain, pleural reactions, cough, and skin burns.

SECONDARY OUTCOMES:
changes of the size about the tumor on CT/MRI images | After the procedures up to three months
  Changes in imaging findings in the ablation zone

CONTACTS AND LOCATIONS:
Overall Officials: Yueyong Xiao, Principal Investigator — The Chinese PLA General Hospital
Locations (1):
- The Chinese PLA General Hospital, Beijing, China